CLINICAL TRIAL: NCT04735458
Title: Investigating Inhibitory Control Networks in Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, J. Nicole Bentley, Principle Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB300003605; 1K23NS117735-01A1 (NIH)
Record Dates: First submitted 2021-01-28; First posted 2021-02-03 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Parkinson's Disease Patients receiving DBS electrodes
  Interventions: Other: Procedure/Surgery: Response Inhibition and Deep Brain Stimulation in Parkinson's disease
- Control (No Intervention): Control subjects will be non-Parkinson's Disease patients with essential tremor

INTERVENTIONS:
Other: Procedure/Surgery: Response Inhibition and Deep Brain Stimulation in Parkinson's disease — After creation of the burr hole and prior to DBS electrode placement, 1-2 subdural strip electrodes will be placed anteriorly or posteriorly from the cranial opening. These electrodes are routinely placed using this technique for seizure mapping, with arrays of electrodes (up to 6) being placed around the perimeter of the opening.14 Subdural strips vary in length and contact size (e.g., the 6-contact Ad-Tech strip), and are currently placed predominantly for studies of sensorimotor function,13 including at our institution (IRB-140327003). Placement over prefrontal areas is performed at other institutions.11-13 The DBS surgery will then proceed according to routine practice, and following lead placement in the optimal desired location, the research task paradigm will begin.
  Arms: Treatment

SUMMARY:
The purpose of this study is to investigate the brain activity associated with non-motor symptoms of movement disorders, including Parkinson's disease and essential tremor. These movement disorders commonly have significant non-motor features also, including depression, cognitive impairment, decreased attention, and slower processing speeds. The investigators are interested in the brain activity associated with these symptoms, and perform recordings of the surface of the brain, in addition to the typical recordings the investigators perform, during routine deep brain stimulation (DBS) surgery.

DETAILED DESCRIPTION:
Movement disorders are a prominent cause of disability worldwide. In the United States, it is estimated that more than 4 million people suffer from Parkinson's disease (PD), essential tremor (ET), and dystonia, some of the most prevalent of neurologic disorders. Of these, PD is the most common, and is primarily characterized by tremor, rigidity, and bradykinesia. However, many patients also have prominent non-motor features, including depression and cognitive impairment, with deficiencies in processing speed, memory, attention, and learning. One of the most debilitating cognitive deficiencies is in response inhibition (RI), or the inability to suppress a habitual action. PD patients have significant difficulty with RI, and report its substantial contribution in limiting their quality of life. While some studies show that dopamine can improve this aspect of cognitive function, many patients remain considerably impaired.

RI manifests clinically in many different and important ways, with reduced mental flexibility, task-switching, and concentration. RI may also contribute to motor impairment, with gait dysfunction, falls, and freezing of gait. Unfortunately, these features of PD and RI are less well-studied and lack effective treatment options, necessitating that new treatments be investigated. Deep brain stimulation (DBS), while a highly effective treatment for motor manifestations, is essentially ineffective for, and can even worsen cognition, with few studies currently investigating how different parameters may improve NMS. In an effort to begin addressing these debilitating features of PD, the investigators propose to study RI in patients with movement disorders, and to correlate movement and cognition with underlying neural electrophysiology before and during tasks of motion and response inhibition.

During routine DBS surgery, the stimulating electrode is implanted with the aid of intraoperative recordings in the awake state. These routine recordings enable neurologists and neurosurgeons to directly observe neuronal firing in the brain, identifying characteristic patterns to delineate anatomic structures. Once in place, the DBS electrode is tested using stimulation parameters known to be clinically efficacious for motor impairment. This allows acute, intraoperative testing for therapeutic benefit and side effects, and give information for how a patient will respond to the therapy once the cranial electrode is connected to the battery and turned on.

In addition to this routine recording and stimulation, this setting also provides a unique opportunity to study neural electrophysiology, with minimal increased risk. By measuring brain activity in the outer layers (cortex) as well as from the DBS electrode itself, while patients perform various tasks, it is possible to correlate behavioral function and neural activity. Our center, and several others, already have research paradigms in place to achieve these goals, by placing a subdural strip electrode over cortex prior to placing the DBS lead. These strip electrodes lie along the surface of the brain, and have historically been used for several decades to perform seizure mapping, typically as an array of electrodes placed via a burr hole. Their use has only more recently been implemented for investigation of neural circuits during DBS surgery, however, their safety in this specific setting is now well-established, and their temporary placement is currently being performed in similar studies at this institution. However, though previous studies have placed these strips over prefrontal areas, the vast majority of research in this area is focused on motor circuits, with placement over sensorimotor cortex. In order to study NMS, strips will be placed over prefrontal cortex, with recordings made during various motor and cognitive tasks and during different stimulation patterns.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for surgery based on multi-disciplinary consensus review
* Have a diagnosis of Parkinson's disease or Essential Tremor
* Have a diagnosis of medically-refractory movement disorder (Parkinson's disease, Essential Tremor, or dystonia)
* Willingness to participate in the paradigms described in the protocol

Exclusion Criteria:

* Inability to provide full and informed consent
* Age younger than 18
* Are not able to participate in study-related activities
* History of prior ischemic/hemorrhagic stroke, subdural hemorrhage, or seizure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy via Simon Task (% correct) | Baseline
  In the Simon task, participants are instructed to respond with a right or left button press (Right = Red, Left = Blue) according to how a word is printed on a screen ("RED" or "BLUE"), regardless of the color in which the word is printed.
  This is a measurement of accuracy (% correct, ranging from 0-100, with higher scores indicating better performance)
Response times via Simon Task (sec) | Baseline
  In the Simon task, participants are instructed to respond with a right or left button press according to the word "RIGHT" or "LEFT" that appears on a screen, regardless of where on the screen it actually appears.
  This is a measurement response times (continuous measure, from 0-4000 milliseconds) between correct and incorrect responses.
Simon Effect on Response times (sec) | Baseline
  Participants will perform the Simon task as described, and the Simon effect will be calculated as the difference in response times between congruent and incongruent trials
Simon Effect on Accuracy (% correct) | Baseline
  Participants will perform the Simon task as described, and the Simon effect will be calculated as the difference in accuracy between congruent and incongruent trials
United Parkinson's disease Rating Scale part 3: Motor Examination Score 0-108 (Higher score represents worse symptoms) | Baseline
  Participants will undergo motor evaluation using the validated United Parkinson's disease Rating Scale (UPDRS) part 3.
Dementia Rating Scale Score 0-144 points (Higher score represents better symptoms) | Baseline
  Participants will undergo neuropsychological testing as part of routine care, including the Dementia Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Bentley, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States